CLINICAL TRIAL: NCT07353008
Title: Effect of Different Chelation Protocols on the Healing of Periapical Lesions in Teeth With Chronic Apical Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Merve Sari, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2801
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Apical Periodontitis
Keywords: Etidronic acid (HEBP); Ethylenediaminetetraacetic acid (EDTA); Sequential chelation; Consecutive chelation
MeSH Terms: interventions — Edetic Acid; Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, parallel-group, double-blind, randomized controlled clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: Final irrigation with 2.5% NaOCl and 17% EDTA (Active Comparator): After preparation of the access cavity the working length (WL) will be determined using an electronic apex locator (Root ZX [Morita, Tokyo, Japan]) and confirmed radiographically. Following glide path preparation, the root canals will be shaped to the working length using a Resiproc files (VDW, Munich, Germany) in accordance with the manufacturer's instructions, employing the crown-down preparation technique.
  During canal preparation, irrigation will be performed with a total of 20 mL of 2.5% NaOCl. After completion of preparation, irrigation will be carried out with 10 mL of distilled water, followed by sequential irrigation with 3 mL of 17% EDTA, 10 mL of distilled water, and 2 mL of 2.5% NaOCl.
  Interventions: Procedure: Final irrigation with 2.5% NaOCl and 17% EDTA
- Group II: Final irrigation with 2.5% NaOCl and 9% HEBP (Experimental): After preparation of the access cavity, the working length (WL) will be determined using an electronic apex locator (Root ZX [Morita, Tokyo, Japan]) and confirmed radiographically. Following glide path preparation, the root canals will be shaped to the working length using a Resiproc files (VDW, Munich, Germany) in accordance with the manufacturer's instructions, employing the crown-down preparation technique.
  During canal preparation, irrigation will be performed with a total of 20 mL of 2.5% NaOCl. After completion of preparation, irrigation will be carried out with 10 mL of distilled water, followed by final irrigation with 5 mL of 2.5% NaOCl-9% HEBP.
  Interventions: Procedure: Final irrigation with 2.5% NaOCl and 9% HEBP
- Group III: Irrigation with 2.5% NaOCl-9% HEBP during both preparation and final irrigation (Experimental): After preparation of the access cavity, the working length (WL) will be determined using an electronic apex locator (Root ZX [Morita, Tokyo, Japan]) and confirmed radiographically. Following glide path preparation, the root canals will be shaped to the working length using a Resiproc files (VDW, Munich, Germany) in accordance with the manufacturer's instructions, employing the crown-down preparation technique.
  During both canal preparation and final irrigation, a total of 25 mL of 2.5% NaOCl-9% HEBP will be used for irrigation.
  Interventions: Procedure: Irrigation with 2.5% NaOCl-9% HEBP during both preparation and final irrigation

INTERVENTIONS:
Procedure: Final irrigation with 2.5% NaOCl and 17% EDTA — During canal preparation, irrigation will be performed with a total of 20 mL of 2.5% NaOCl. After completion of preparation, irrigation will be carried out with 10 mL of distilled water, followed by sequential irrigation with 3 mL of 17% EDTA, 10 mL of distilled water, and 2 mL of 2.5% NaOCl.
  Arms: Group I: Final irrigation with 2.5% NaOCl and 17% EDTA
Procedure: Final irrigation with 2.5% NaOCl and 9% HEBP — During canal preparation, irrigation will be performed with a total of 20 mL of 2.5% NaOCl. After completion of preparation, irrigation will be carried out with 10 mL of distilled water, followed by final irrigation with 5 mL of 2.5% NaOCl-9% HEBP.
  Arms: Group II: Final irrigation with 2.5% NaOCl and 9% HEBP
Procedure: Irrigation with 2.5% NaOCl-9% HEBP during both preparation and final irrigation — During both canal preparation and final irrigation, a total of 25 mL of 2.5% NaOCl-9% HEBP will be used for irrigation.
  Arms: Group III: Irrigation with 2.5% NaOCl-9% HEBP during both preparation and final irrigation

SUMMARY:
The aim of this study is to evaluate the effects of different irrigation protocols using ethylenediaminetetraacetic acid (EDTA) and etidronic acid (HEBP) on periapical lesion healing and postoperative pain in single-rooted, single-canal mandibular anterior and premolar teeth diagnosed with chronic apical periodontitis.

DETAILED DESCRIPTION:
Materials and Methods Study Design This study was designed as a randomized clinical trial with three parallel experimental arms and included data obtained from a total of 63 patients.

Randomization and Blinding

Patients were randomly allocated to one of the following three groups:

Irrigation with 2.5% sodium hypochlorite (NaOCl) during canal preparation and 17% ethylenediaminetetraacetic acid (EDTA) as the final irrigant; Irrigation with 2.5% NaOCl during canal preparation and a combination of 2.5% NaOCl and 9% etidronic acid (HEBP) as the final irrigant; Irrigation with a mixture of 2.5% NaOCl and 9% HEBP throughout the entire irrigation protocol.

Randomization was performed using an online randomization tool (www.randomizer.org). Block randomization with a block size of four was applied to ensure an equal 1:1 allocation among the study groups. All endodontic procedures were performed by a single experienced operator. Due to the inherent differences between the irrigation protocols, blinding of the patients, the operator, and the radiographic evaluator was not feasible.

Clinical Intervention Inferior alveolar nerve block anesthesia was administered using 4% articaine with 1:100,000 epinephrine (Ultracain DS; Sanofi-Aventis, Germany). Following rubber dam isolation, all carious tissue was removed non-selectively under water cooling using a sterile high-speed diamond bur, and cavity preparation was completed with a sterile round bur mounted on a low-speed handpiece.

Subsequently, root canal treatment was performed according to the assigned group protocol, consisting of either 2.5% NaOCl and 17% EDTA as the final irrigation regimen, 2.5% NaOCl and 9% HEBP as the final irrigation regimen, or 2.5% NaOCl and 9% HEBP used both during canal preparation and as the final irrigation solution.

Irrigation Procedures Group I: Final Irrigation with 2.5% NaOCl and 17% EDTA After access cavity preparation, the working length (WL) was determined using an electronic apex locator (Root ZX; Morita, Tokyo, Japan) and confirmed radiographically. Following glide path preparation, the root canals were shaped to the working length using Reciproc files (VDW, Munich, Germany) according to the manufacturer's instructions, employing a crown-down preparation technique. During canal instrumentation, irrigation was performed with a total volume of 20 mL of 2.5% NaOCl. Upon completion of canal preparation, irrigation was carried out sequentially with 10 mL of distilled water, 3 mL of 17% EDTA, 10 mL of distilled water, and a final rinse with 2 mL of 2.5% NaOCl.

Group II: Final Irrigation with 2.5% NaOCl and 9% HEBP After access cavity preparation, the working length was determined using an electronic apex locator and confirmed radiographically. Following glide path preparation, root canal shaping was performed to the working length using Reciproc files in accordance with the manufacturer's recommendations and a crown-down technique. During canal preparation, irrigation was performed using a total of 20 mL of 2.5% NaOCl. After instrumentation, the canals were irrigated with 10 mL of distilled water, followed by final irrigation with 5 mL of a solution containing 2.5% NaOCl and 9% HEBP.

Group III: Irrigation with 2.5% NaOCl-9% HEBP During Both Preparation and Final Irrigation After access cavity preparation, the working length was established using an electronic apex locator and confirmed radiographically. Glide path preparation was followed by canal shaping to the working length using Reciproc files with a crown-down technique. Throughout both canal preparation and final irrigation, a total of 25 mL of a solution containing 2.5% NaOCl and 9% HEBP was used for irrigation.

Root Canal Obturation Following completion of the irrigation procedures, the root canals were dried with sterile paper points and obturated using gutta-percha cones in combination with a calcium silicate-based sealer, employing the cold lateral condensation technique. A postoperative periapical radiograph was obtained after obturation. Teeth exhibiting overfilling beyond the radiographic apex or obturation terminating more than 2 mm short of the apex were excluded from the study.

Final Restoration A 3-mm-thick layer of flowable composite resin was placed in the pulp chamber. The remaining coronal restoration was completed using composite resin with an incremental layering technique. After removal of the rubber dam, occlusal adjustments were performed, and the restoration was finished and polished during the same appointment. Immediate postoperative periapical radiographs were then obtained.

Patients were instructed to return for follow-up examinations at 3, 6, and 12 months, or earlier if any symptoms occurred.

Postoperative Pain Management For postoperative pain control, patients were prescribed 400 mg ibuprofen tablets to be taken as needed. Patients were instructed to record the frequency of analgesic intake in writing. In cases of severe postoperative pain not relieved by analgesics, patients were advised to contact the operator immediately.

Evaluation Criteria and Follow-up Examinations Clinical and Radiographic Follow-up Patients were recalled at 3, 6, and 12 months for clinical and radiographic examinations. At each follow-up visit, the clinical and radiographic outcomes of the treated teeth were recorded.

Clinical Success Criteria

Clinical success was defined as:

Absence of spontaneous pain or discomfort, except during the initial postoperative days; Absence of tooth mobility greater than Grade I; Normal periradicular soft tissues without swelling or sinus tract formation; Negative responses to axial palpation and percussion tests. Radiographic Success Criteria

Radiographic success was defined as:

No increase in the Periapical Index (PAI) score at follow-up; Absence of extra-radicular or intra-radicular pathology; No evidence of internal or external root resorption. Additional Assessments The integrity of the coronal restoration was evaluated at each follow-up visit, and any need for replacement or re-restoration was recorded. Additionally, the presence of clinical symptoms, including percussion sensitivity, sinus tract formation, and extraoral abscess, was assessed at all follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients of both sexes aged 18-60 years, with no systemic diseases, will be screened for inclusion in the study. Strict eligibility criteria will be applied.

Eligible patients will present with restorable mandibular single-rooted premolar and anterior teeth, a healthy periodontal status (periodontal pocket depth ≤3 mm), and a clinical diagnosis of chronic apical periodontitis. The diagnosis of chronic apical periodontitis will be based on the absence of clinical symptoms, the presence of pulpal necrosis, negative responses to electric pulp testing and cold testing, and the detection of a radiolucent area in the periapical region on radiographic examination. In addition, included teeth must exhibit a periapical lesion with a Periapical Index (PAI) score of 2 or higher.

Exclusion Criteria:

* Patients with systemic diseases (such as diabetes mellitus, hypertension, chronic liver disease, or coagulation disorders), those with bone metabolism disorders and/or those using medications that affect bone metabolism (including steroids and bisphosphonates), and pregnant patients will be excluded from the study.

In addition, teeth presenting with periodontal pocket depths greater than 3 mm, internal or external root resorption, vertical or horizontal root fractures, a history of previous root canal treatment, the presence of a sinus tract, or intraoral or extraoral abscess associated with the involved tooth, as well as teeth deemed non-restorable, will not be included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Periapical Lesion Healing | 1 year
  Radiographic periapical status assessed using the Periapical Index (PAI) according to Ørstavik et al., with scores ranging from 1 (normal periapical structures) to 5 (severe apical periodontitis), based on the degree of periapical radiolucency. The primary outcome will be periapical lesion healing, evaluated by changes in periapical index (PAI) scores on periapical radiographs taken before treatment and at the 12-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endodontics, Faculty of Dentistry, Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD due to confidentiality and privacy considerations.

REFERENCES:
- [Result] Campello AF, Rodrigues RCV, Alves FRF, Miranda KR, Brum SC, Mdala I, Siqueira JF Jr, Rocas IN. Enhancing the Intracanal Antibacterial Effects of Sodium Hypochlorite with Etidronic Acid or Citric Acid. J Endod. 2022 Sep;48(9):1161-1168. doi: 10.1016/j.joen.2022.06.006. Epub 2022 Jun 22. PMID 35750221
- [Result] Hazar E, Hazar A. Effects of phytic acid and etidronic acid using continuous and sequential chelation on the removal of smear layer, dentin microhardness, and push-out bond strength of calcium silicate-based cement. BMC Oral Health. 2025 Apr 24;25(1):633. doi: 10.1186/s12903-025-06010-5. PMID 40275217
- [Result] Tartari T, Wilchenski BS, de Souza Lima LA, Vivan RR, Ballal V, Duarte MAH. The use of sodium hypochlorite mixed with etidronic acid during canal preparation increases debris extrusion. Aust Endod J. 2023 Dec;49(3):584-591. doi: 10.1111/aej.12788. Epub 2023 Aug 11. PMID 37571801
- [Result] Razumova S, Brago A, Kryuchkova A, Troitskiy V, Bragunova R, Barakat H. Evaluation of the efficiency of smear layer removal during endodontic treatment using scanning electron microscopy: an in vitro study. BMC Oral Health. 2025 Jan 28;25(1):151. doi: 10.1186/s12903-025-05510-8. PMID 39875846
- [Result] Pandya DS, Kritika S, Sanjeev K, Mahalaxmi S, Neelakantan P. Endotoxin Levels after Calcium Hydroxide Placement in Root Canals Irrigated with Continuous or Sequential Chelation in Previously Treated Teeth with Symptomatic Apical Periodontitis: A Randomized Controlled Clinical Trial. J Endod. 2025 Nov;51(11):1519-1525. doi: 10.1016/j.joen.2025.08.004. Epub 2025 Aug 18. PMID 40835176